CLINICAL TRIAL: NCT01370512
Title: Treatment Trial of Droxidopa and Pyridostigmine to Improve Orthostatic Hypotension Without Aggravating Supine Hypertension
Brief Title: Droxidopa / Pyridostigmine in Orthostatic Hypotension
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Wolfgang Singer, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-008810; P01NS044233 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic | interventions — Droxidopa; Pyridostigmine Bromide

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind, randomized four-way crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo, Then Pyridostigmine (Active Comparator): participants first receive placebo by mouth 3 times a day, for treatment day 1. Then participants receive pyridostigmine by mouth 3 times a day for treatment day 2.
  Interventions: Drug: Pyridostigmine; Other: Placebo
- Pyridostigmine, Then Placebo (Active Comparator): participants first receive pyridostigmine by mouth 3 times a day, for treatment day 1. Then participants receive placebo by mouth 3 times a day for treatment day 2.
  Interventions: Drug: Pyridostigmine; Other: Placebo
- Drioxidopa and Placebo, Then Drioxidopa and Pyridostigmine (Experimental): participants first receive placebo by mouth 3 times a day, for treatment day 3. Then participants receive Droxidopa by mouth 3 times a day for treatment day 4.
  Interventions: Drug: Droxidopa; Drug: Pyridostigmine; Other: Placebo
- Droxidopa and Pyridostigmine, Then Droxidopa and Placebo (Experimental): participants first receive Droxidopa by mouth 3 times a day, for treatment day 3. Then participants receive Placebo by mouth 3 times a day for treatment day 4.
  Interventions: Drug: Droxidopa; Drug: Pyridostigmine; Other: Placebo

INTERVENTIONS:
Drug: Droxidopa — 100 mg tablets by mouth three times a day
  Arms: Drioxidopa and Placebo, Then Drioxidopa and Pyridostigmine; Droxidopa and Pyridostigmine, Then Droxidopa and Placebo
Drug: Pyridostigmine — 60 mg tablets by mouth three times a day
Other: Placebo — Looks exactly like the study drug but contains no active ingredients

SUMMARY:
This study is being done to study the combination of pyridostigmine and low-dose Droxidopa for the treatment of orthostatic hypotension.

ELIGIBILITY:
Inclusion Criteria

1. The presence of OH (fall in systolic BP >=30 mm Hg) is required for this study.
2. Autonomic testing and clinical evaluation demonstrates OH to be of neurogenic etiology.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Chronic illnesses or the presence of other conditions that potentially involve the CNS or affect autonomic testing. These include congestive heart failure, recent (<6 months) myocardial infarct, severe anemia, diabetes mellitus, alcoholism, malignant neoplasms, amyloidosis, hypothyroidism, sympathectomy, cerebrovascular accidents, and neurotoxins or neuroactive drug exposure.
3. Orthopedic problems or cardiopulmonary disease, sufficient to compromise mobility and activity of daily living.
4. Any known concurrent infection or severe liver or kidney disease.
5. Medications that could affect autonomic function are suspended prior to autonomic testing. Therapy with midodrine, alpha and beta adrenergic antagonists, or other medications that affect autonomic function will be withdrawn 48 hours prior to autonomic evaluations. Fludrocortisone doses up to 0.2 mg per day will be permitted. Stable doses of antidepressants (tricyclics, SSRIs, SNRIs) will also be permitted. The 48h medication withdrawal is reviewed on a case by case basis - if felt unsafe by the investigators, the withdrawal period may be shortened. This will be documented in the study documents.
6. Occasional use of a neuroleptic as an anti-emetic in the past is allowed, but none can have been used within 3 weeks prior to this study.
7. Use of methylphenidate, cinnarizine, reserpine, amphetamine, atypical antipsychotics such as risperidone, olanzapine, and quetiapine or a MAO-A inhibitor within 3 weeks prior to this study.
8. Dementia (DSM-IV criteria - Amer. Psych. Assoc., 1994). The score on the Mini-Mental State Examination must be >24.
9. History of stroke (diagnosed on clinical grounds as an acute deterioration of neurological function typical of a stroke; confirmatory CT or MRI evidence of stroke will be useful but not necessary).
10. History of electroconvulsive therapy.
11. History of brain surgery for Parkinson's disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in orthostatic diastolic blood pressure | 1 hour after medication administration, 2 hours after medication administration
  diastolic blood pressure measured upon standing reported in mm/Hg

SECONDARY OUTCOMES:
Change in orthostatic systolic blood pressure | 1 hour after medication administration, 2 hours after medication administration
  systolic blood pressure measured upon standing reported in mm/Hg
Change in absolute supine diastolic blood pressure | 1 hour after medication administration, 2 hours after medication administration
  diastolic blood pressure measured while lying flat reported in mm/Hg
Change in absolute supine systolic blood pressure | 1 hour after medication administration, 2 hours after medication administration
  systolic blood pressure measured while lying flat reported in mm/Hg
Change in supine norepinephrine levels | 1 hour after medication administration, 2 hours after medication administration
  measure of serum norepinephrine levels while lying flat reported in pg/mL
Change in orthostatic symptoms | 1 hour after medication administration, 2 hours after medication administration
  measured during tilt study, the patient will be asked to score orthostatic symptoms on a symptom scale ranging from "0" = no symptoms to "10" = near syncope

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Singer, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No